CLINICAL TRIAL: NCT05602194
Title: A Randomized Trial of Levocarnitine Prophylaxis to Prevent Asparaginase-Associated Hepatotoxicity in Adolescents and Young Adults Receiving Acute Lymphoblastic Leukemia Therapy
Brief Title: Studying the Effect of Levocarnitine in Protecting the Liver From Chemotherapy for Leukemia or Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACCL1931; NCI-2022-08058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL1931 (Other: Children's Oncology Group); COG-ACCL1931 (Other: DCP); ACCL1931 (Other: CTEP); U24CA196173 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2022-10-18; First posted 2022-11-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: B Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; B Acute Lymphoblastic Leukemia, BCR-ABL1-Like; Lymphoblastic Lymphoma; Mixed Phenotype Acute Leukemia; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; calaspargase pegol; Asparaginase; Carnitine; pegaspargase

STUDY DESIGN:
Intervention Model Description: Parallel with the option to cross over to Arm C to begin levocarnitine rescue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (levocarnitine, standard of care chemotherapy) (Experimental): Patients receive levocarnitine PO or IV as a bolus over 2 to 3 minutes or by infusion (over 10 to 30 minutes or per institutional standard) starting prior to standard of care induction chemotherapy with pegaspargase or calaspargase pegol and continued through the earlier of the last day of Induction phase (i.e., day prior to start of next phase) or Induction day 35. Patients may also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Calaspargase Pegol; Dietary Supplement: Levocarnitine; Drug: Pegaspargase; Other: Quality-of-Life Assessment
- Arm B (standard of care chemotherapy) (Active Comparator): Patients receive standard of care induction chemotherapy with pegaspargase or calaspargase pegol on study. Patients may also undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Calaspargase Pegol; Drug: Pegaspargase; Other: Quality-of-Life Assessment
- Arm C (rescue levocarnitine) (Experimental): Patients in Arms A and B who develop conjugated hyperbilirubinemia > 3 mg/dL during induction may receive levocarnitine rescue PO or IV as a bolus dose over 2 to 3 minutes or by infusion (over 10 to 30 minutes or per institutional standard) until resolution of conjugated hyperbilirubinemia =< 3 mg/dL (or start of consolidation or the next treatment phase, whichever occurs first).
  Interventions: Dietary Supplement: Levocarnitine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm A (levocarnitine, standard of care chemotherapy); Arm B (standard of care chemotherapy)
Drug: Calaspargase Pegol — Given standard of care calaspargase pegol
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Arm A (levocarnitine, standard of care chemotherapy); Arm B (standard of care chemotherapy)
Dietary Supplement: Levocarnitine — Given PO or IV
  Other Names: Carnitor; L-carnitine
  Arms: Arm A (levocarnitine, standard of care chemotherapy); Arm C (rescue levocarnitine)
Drug: Pegaspargase — Given standard of care pegaspargase
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Arm A (levocarnitine, standard of care chemotherapy); Arm B (standard of care chemotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm A (levocarnitine, standard of care chemotherapy); Arm B (standard of care chemotherapy)

SUMMARY:
This phase III trial compares the effect of adding levocarnitine to standard chemotherapy versus (vs.) standard chemotherapy alone in protecting the liver in patients with leukemia or lymphoma. Asparaginase is part of the standard of care chemotherapy for the treatment of acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma (LL), and mixed phenotype acute leukemia (MPAL). However, in adolescent and young adults (AYA) ages 15-39 years, liver toxicity from asparaginase is common and often prevents delivery of planned chemotherapy, thereby potentially compromising outcomes. Some groups of people may also be at higher risk for liver damage due to the presence of fat in the liver even before starting chemotherapy. Patients who are of Japanese descent, Native Hawaiian, Hispanic or Latinx may be at greater risk for liver damage from chemotherapy for this reason. Carnitine is a naturally occurring nutrient that is part of a typical diet and is also made by the body. Carnitine is necessary for metabolism and its deficiency or absence is associated with liver and other organ damage. Levocarnitine is a drug used to provide extra carnitine. Laboratory and real-world usage of the dietary supplement levocarnitine suggests its potential to prevent or reduce liver toxicity from asparaginase. The overall goal of this study is to determine whether adding levocarnitine to standard of care chemotherapy will reduce the chance of developing severe liver damage from asparaginase chemotherapy in ALL, LL and/or MPAL patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine in a randomized manner whether the addition of levocarnitine prophylaxis to asparaginase-containing regimens will decrease the incidence of conjugated hyperbilirubinemia (> 3 mg/dL) during ALL induction therapy for adolescents and young adults (adolescents and young adults [AYAs], age 15-39 years).

SECONDARY OBJECTIVES:

I. To examine the impact of levocarnitine prophylaxis on differences in the incidence of grade >= 3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations during ALL Induction.

II. To compare rates of minimal residual disease (MRD) positivity at end of Induction and describe MRD+ by end of consolidation (EOC) in those receiving ALL induction chemotherapy with and without levocarnitine.

EXPLORATORY OBJECTIVES:

I. To compare rates of toxicity and associated dose reductions for chemotherapy administered with and without concomitant levocarnitine supplementation.

II. To compare across study arms the peak levels during Induction of conjugated and total bilirubin, AST, ALT, and duration of conjugated hyperbilirubinemia from onset > 3 mg/dL to =< 3 mg/dL.

III. To describe the efficacy of levocarnitine prophylaxis to reduce the incidence and/or severity of early patient-reported chemotherapy-induced peripheral neuropathy.

IV. To describe the three-year event-free and overall survival (EFS/OS) in those treated with and without levocarnitine prophylaxis.

V. To examine the association of age with asparaginase activity and asparaginase-associated hepatotoxicity during induction.

VI. To examine the association of body-mass-index (BMI) percentile (or absolute BMI for young adults) with asparaginase activity and asparaginase-associated hepatotoxicity during induction.

VII. To describe adherence by self-report and pill-count to oral levocarnitine in patients randomized to the intervention arm.

VIII. To examine the association of plasma levels of carnitine and related markers with the efficacy of levocarnitine supplementation.

IX. To determine the impact of inherited genetic variation on hepatoxicity and levocarnitine efficacy.

OUTLINE: Patients are randomized to 1 of 2 arms (arm A vs. B).

ARM A: Patients receive levocarnitine orally (PO) or intravenously (IV) as a bolus over 2 to 3 minutes or by infusion (over 10 to 30 minutes or per institutional standard) starting prior to standard of care induction chemotherapy with pegaspargase or calaspargase pegol and continued through the earlier of the last day of Induction phase (i.e., day prior to start of next phase) or Induction day 35. Patients may also undergo blood sample collection during screening and on study.

ARM B: Patients receive standard of care induction chemotherapy with pegaspargase or calaspargase pegol on study. Patients may also undergo blood sample collection during screening and on study.

ARM C (RESCUE): Patients in Arms A and B who develop conjugated hyperbilirubinemia > 3 mg/dL during induction may receive levocarnitine rescue PO or IV as a bolus dose over 2 to 3 minutes or by infusion (over 10 to 30 minutes or per institutional standard) until resolution of conjugated hyperbilirubinemia =< 3 mg/dL (or start of consolidation or the next treatment phase, whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* >= 15 and < 40 years at time of diagnosis
* Newly diagnosed B-ALL, T-ALL, lymphoblastic lymphoma (LLy), or mixed-phenotype acute leukemia/lymphoma (MPAL)

  * Note: Philadelphia chromosome (PH)+ and PH-like acute leukemia are eligible (use of tyrosine kinase inhibitors [TKI] or CRLF2- targeted concomitant medication must be documented, if used)
* Conjugated bilirubin =< 1.5 x upper limit of normal (ULN) for age, regardless of baseline bilirubin (within 7 days prior to enrollment), and
* Serum glutamate pyruvate transaminase (SGPT) (ALT) =< 225 U/L (=< 5x ULN) (within 7 days prior to enrollment), and

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L and serum glutamic oxaloacetic transaminase (SGOT) (AST) to 50 U/L regardless of baseline
* SGOT (AST) =< 250 U/L (=< 5x ULN) (within 7 days prior to enrollment)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L and SGOT (AST) to 50 U/L regardless of baseline
* For patients receiving ursodiol prior to enrollment, laboratory values must meet above criteria off ursodiol for 7 days
* PEDIATRIC PATIENTS (AGE 15-17 years):

  * A 24-hour urine creatinine clearance >= 30 mL/min/1.73 m^2 (within 7 days prior to enrollment) OR
  * A glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2. GFR must be performed using one of the following methods (within 7 days prior to enrollment):

    * 1. Estimated GFR (eGFR) >= 30 mL/min/1.73 m^2.

      * An online calculator is available through the National Kidney Foundation at https://www.kidney.org/professionals/kdoqi/gfr_calculatorped
    * 2. Measured GFR >= 30 mL/min/1.73 m^2 (any age). If measured GFR is used, it must be performed using direct measurement with a nuclear blood sampling method or small molecule clearance method (iothalamate or other molecule per institutional standard).
* ADULT PATIENTS (AGE 18 YEARS OR OLDER): Creatinine clearance >= 30 mL/min, as estimated by the Cockcroft and Gault formula or a 24-hour urine collection (within 7 days prior to enrollment). Estimated creatinine clearance is based on actual body weight

  * An online calculator is available through the National Kidney Foundation at https://www.kidney.org/professionals/kdoqi/gfr_calculatorcoc
* Berlin-Frankfurt-Munich (BFM), Children's Oncology Group (COG), or C10403-based Induction regimen and must be inclusive of >= 1 dose of pegaspargase or calaspargase pegol, and
* First dose of asparaginase must be planned within the first week of induction therapy, and
* Dose of pegaspargase or calaspargase pegol must be >= 1,000 IU/ m^2 (dose-capping permitted per primary regimen)

  * Note: Co-enrollment on a therapeutic consortia trial is not required
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Down syndrome
* Known inherited or autoimmune liver disease impacting conjugated bilirubin (e.g., Alagille syndrome, primary sclerosing cholangitis, other)
* Known biopsy (or imaging) proven severe liver fibrosis (Batts-Ludwig >= stage 3)
* Unable to tolerate oral formulation of study drug at enrollment
* Patients who received chemotherapy or treatment for a prior malignancy are not eligible

  * The following are permitted: steroid prophase, hydroxyurea, or other cytoreduction prior to initiation of Induction chemotherapy (must be documented) and chemotherapy for current diagnosis (i.e. initiation of Induction therapy within enrollment window). Chemotherapy prior to enrollment for treatment of a non-malignancy (e.g., steroid or methotrexate for autoimmune disease) is also permitted and must be documented
* Female patients who are pregnant since fetal toxicities and teratogenic effects in humans are unknown for study drug. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of conjugated hyperbilirubinemia >3 mg/dL during induction therapy | During induction therapy (up-to 35-days after initiating induction chemotherapy)
  For patients assigned to arms A and B, the investigators will separately estimate the proportion of patients who experience conjugated hyperbilirubinemia > 3mg/dL during induction chemotherapy by arm along with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of grade >= 3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations during induction therapy | During induction therapy (up-to 35-days after initiating induction chemotherapy)
  For patients assigned to arms A and B, the investigators will separately estimate the proportion of patients who experience grade >= 3 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations during induction chemotherapy by arm along with corresponding 95% confidence intervals.
Incidence of minimal residual disease (MRD) positivity (MRD >= 0.01%) | At end of induction chemotherapy (up-to 35-days after initiating induction chemotherapy), and at end of consolidation chemotherapy (up-to day 56 days after initiating induction chemotherapy)
  For patients assigned to arms A and B, the proportion having MRD positivity at the end of induction chemotherapy will be estimated separately by arm along with corresponding 95% confidence intervals. For patients assigned to arms A and B, the proportion having MRD positivity at the end of consolidation chemotherapy will be estimated separately by arm along with corresponding 95% confidence intervals (only patients with end of consolidation MRD evaluated and who did not get placed on the rescue arm C will be included).

OTHER OUTCOMES:
Incidence of Common Terminology Criteria for Adverse Events (CTCAE) grade >= 4 adverse events during induction chemotherapy | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the proportion experiencing CTCAE grade >=4 adverse events by the end of induction chemotherapy will be estimated along with 95% confidence intervals.
Incidence of daunorubicin, vincristine, and/or asparaginase chemotherapy dose reductions during induction chemotherapy | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the proportion receiving a dose reduction during induction chemotherapy relative to planned doses at the beginning of induction chemotherapy for daunorubicin, vincristine, and/or asparaginase will be estimated along with 95% confidence intervals
Percentage of planned dose given for daunorubicin, vincristine, and/or asparaginase during induction chemotherapy | Up to 35 days (induction phase)
  For patients assigned to arms A and b, the median percent planned dose given during induction will also be calculated as well as 95% confidence intervals.
Peak levels during induction of conjugated bilirubin | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the investigators will calculate median peak conjugated bilirubin as well as corresponding 95% confidence intervals.
Peak levels during induction of total bilirubin | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the investigators will calculate median peak ALT as well as corresponding 95% confidence intervals.
Peak levels of AST during induction chemotherapy | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the investigators will calculate median peak ALT as well as corresponding 95% confidence intervals.
Peak levels of ALT during induction chemotherapy | Up to 35 days (induction phase)
  For patients assigned to arms A and B, the investigators will calculate median peak ALT as well as corresponding 95% confidence intervals.
Days of conjugated hyperbilirubinemia (> 3 mg/dL) to <=3 mg/dL during induction | Up to 35 days (induction phase)
  For patients assigned to arms A, B, and C, the investigators will calculate the median days from onset of conjugated hyperbilirubinemia as well as 95% confidence intervals.
Severity of patient-reported chemotherapy induced peripheral neuropathy (CIPN) as measured by the 11-question Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) survey | Up to 35 days (induction phase)
  The 11-question FACT/GOG-NTX survey will be used to assess patient reported CIPN, where a higher score indicates more severe CIPN. For patients on arms A and B, a median and corresponding 95% confidence interval will be estimated and reported.
Event free survival (EFS) | The time from randomization to first event (relapse, second malignant neoplasm, remission or death) or date of last contact for those who are disease-free, assessed up to 3 years
  For EFS analysis, 3-year EFS probabilities and corresponding 95% confidence interval (CI) will be estimated for Arms A and B, separately, using the Kaplan Meier method. A log-rank test will be used to compare EFS between Arm A versus Arm B (Arm C patients will not contribute to this analysis after they start levocarnitine rescue). Additional EFS analyses comparing Arms A versus B will also be performed using Cox regression models adjusted for "levocarnitine rescue" (i.e., Arm C patients/time) as a time-varying covariate. Hazard ratio and the corresponding 95%CI will be reported for each arm.
Overall survival (OS) | Time from study entry to death or date of last contact for those alive at last contact, assessed up to 3 years
  For OS analysis, 3-year OS probabilities and corresponding 95% CI will be estimated for Arms A and B, separately, using the Kaplan Meier method.
Asparaginase activity | Days 8, 15, and 22
  Spearman's correlation coefficients and corresponding 95% confidence intervals will be reported comparing asparaginase activity to age and BMI.
Association of body-mass-index (BMI) percentile (or absolute BMI for young adults) with asparaginase activity and asparaginase-associated hepatotoxicity during induction therapy | Days 8, 15, and 22
  The association of BMI percentile with asparaginase activity will be assessed using Spearman's correlation. Logistic regression will be used to separately assess the relationship of BMI (considered as a continuous variable and an ordinal variable) and asparaginase activity with hepatotoxicity (conjugated hyperbilirubinemia, ALT) dichotomized as conjugated hyperbilirubinemia >3 versus =< 3 mg/dl and CTCAE grade >= 3 versus < 3 AST or ALT, respectively. Analyses will be performed separately for asparaginase activity measured on Days ~8, 15, and 22 and for Arms A and B.
Adherence to oral levocarnitine during induction chemotherapy measured by percentage of pills returned relative to those prescribed | Up to 35 days (induction phase)
  Descriptive statistics (mean (sd) or median (range) as appropriate) will be used to summarize adherence to levocarnitine tablets during induction in AYA patients randomized to the intervention Arm A as assessed by self-report (% doses compliant) and pill-counts (% pills returned). The percentage of doses compliant will be calculated as: the number of reported missed doses / total prescribed doses for the entire induction period. And the percentage of pills returned will be calculated as the number of pills returned / (number of pills dispensed - number of pills prescribed not taken [i.e., for prescribed dose reductions for toxicity for the entire induction period]).
Adherence to oral levocarnitine measured by percentage dose compliance (% doses reported taken relative to prescribed) | Up to 35 days (induction phase)
  The investigators will report the median percentage dose compliance across patients assigned to arm A as well as a 95% confidence interval.
Mean plasma levels of carnitine | Up to 3 years
  The Investigators will calculate mean plasma levels of carnitine at baseline and at steady state for patients in arms A and B who do and do not experience conjugated hyperbilirubinemia >3 mg/dL and will calculate corresponding 95% confidence intervals.
Impact inherited genetic variation on hepatoxicity and levocarnitine efficacy | Up to 3 years
  This aim will use specimens banked for future research to describe the association of candidate genes (PNPLA3, SOD2, GST family, other) with conjugated hyperbilirubinemia >3 mg/dL and CTCAE Grade ≥3 AST or ALT elevations between treatment arms. Analyses will include ethnic and racial differences, with ancestry determined by self-report and complementary admixture mapping. The association of observed genetic differences with oxidant stress markers (e.g., protein oxidation, lipid peroxidation, total oxidant capacity) pre- and post-asparaginase will be assessed. In general, a multivariable logistic regression model will be used to examine the association between the occurrence of the primary endpoint and the genetic variant of interest, inclusive of covariates: age, obesity, and treatment versus control arm (1:1).

CONTACTS AND LOCATIONS:
Overall Officials: Etan Orgel, Principal Investigator — Children's Oncology Group
Locations (223):
- United States (220):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario